CLINICAL TRIAL: NCT00049504
Title: Nonmyeloablative Hematopoietic Stem Cell Transplantation for Patients With High-Risk Hematologic Malignancies Using Related, HLA-Haploidentical Donors: A Phase II Trial of Combined Immunosuppression Before and After Transplantation
Brief Title: Haploidentical Donor Bone Marrow Transplant in Treating Patients With High-Risk Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1667.00; NCI-2010-00166 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hematopoietic/Lymphoid Cancer; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Myelodysplastic Syndromes; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage II Multiple Myeloma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Childhood Hodgkin Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Childhood Hodgkin Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Hematologic Neoplasms; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Cyclophosphamide; fludarabine phosphate; Tacrolimus; Mycophenolic Acid; Polymerase Chain Reaction; In Situ Hybridization, Fluorescence; Amplified Fragment Length Polymorphism Analysis; Gene Expression Profiling; Whole-Body Irradiation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Treatment (nonmyeloablative HSCT) (Experimental): NONMYELOABLATIVE CONDITIONING: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 1 hour on days -6 and -5. Patients undergo total body irradiation on day -1.
  TRANSPLANTATION: Patients undergo BMT, from an HLA-haploidentical donor, on day 0.
  POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive cyclophosphamide IV over 1 hour on day 3.
  GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: Patients receive tacrolimus IV over 1-2 hours and then tacrolimus PO, once tolerated, on days 4-180, with taper on day 86 in the absence of graft-versus-host disease. Patients also receive mycophenolate mofetil PO three times daily on days 4-35.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: tacrolimus; Drug: mycophenolate mofetil; Genetic: polymerase chain reaction; Genetic: fluorescence in situ hybridization; Genetic: polymorphism analysis; Genetic: gene expression analysis; Radiation: total-body irradiation; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: tacrolimus — Given IV or orally
  Other Names: FK 506; Prograf
Drug: mycophenolate mofetil — Given orally
  Other Names: Cellcept; MMF
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: fluorescence in situ hybridization — Correlative studies
  Other Names: fluorescence in situ hybridization (FISH)
Genetic: polymorphism analysis — Correlative studies
Genetic: gene expression analysis — Correlative studies
Radiation: total-body irradiation — Undergo total-body irradiation
  Other Names: TBI
Procedure: allogeneic bone marrow transplantation — Undergo haploidentical hematopoietic bone marrow transplantation
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo haploidentical hematopoietic bone marrow transplantation

SUMMARY:
This phase II trial studies how well giving fludarabine phosphate, cyclophosphamide, tacrolimus, mycophenolate mofetil and total-body irradiation together with a donor bone marrow transplant works in treating patients with high-risk hematologic cancer. Giving low doses of chemotherapy, such as fludarabine phosphate and cyclophosphamide, and total-body irradiation before a donor bone marrow transplant helps stop the growth of cancer cells by stopping them from dividing or killing them. Giving cyclophosphamide after transplant may also stop the patient's immune system from rejecting the donor's bone marrow stem cells. The donated stem cells may replace the patient's immune system cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and mycophenolate mofetil after the transplant may stop this from happening

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine if engraftment can be achieved safely in patients with high-risk hematologic malignancies who undergo non-myeloablative bone marrow transplantation (BMT) from human leukocyte antigen (HLA)-haploidentical donors.

OUTLINE:

NONMYELOABLATIVE CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) over 1 hour on days -6 to -2 and cyclophosphamide IV over 1 hour on days -6 and -5. Patients undergo total body irradiation on day -1.

TRANSPLANTATION: Patients undergo BMT, from an HLA-haploidentical donor, on day 0.

POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive cyclophosphamide IV over 1 hour on day 3.

GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: Patients receive tacrolimus IV over 1-2 hours and then tacrolimus orally (PO), once tolerated, on days 4-180, with taper on day 86 in the absence of graft-versus-host disease. Patients also receive mycophenolate mofetil PO three times daily on days 4-35.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Chronic myeloid leukemia (CML) in accelerated phase (AP)
* Acute myeloid leukemia (AML) with high-risk cytogenetics [del(5q)/-5, del(7q)/-7, abnormal 3q, 9q, 11q, 20q, 21q, 17p, t(6:9), t(9;22), complex karyotypes (>= 3 abnormalities)] in complete remission (CR)1
* AML >= CR2; patients should have < 5% marrow blasts at the time of transplant
* High-risk ALL defined as: CR1 with high-risk cytogenetics; t(9;22), t(4;11), or hypodiploid (< 45 chromosomes) for pediatric patients; t(9;22), t(8;14), t(4;11), t(1;19) for adult patients; > 4 wk to achieve CR1; >= CR2 (patients should have < 5% marrow blasts at the time of transplant)
* Myelodysplastic syndromes (MDS) (>int-1 per IPSS) after >= 1 prior cycle of induction chemotherapy; should have < 5% marrow blasts at the time of transplant
* Multiple myeloma (MM) Stage II or III patients who have progressed after an initial response to chemotherapy or autologous hematopoietic stem cell transplantation (HSCT) or MM patients with refractory disease who may benefit from tandem autologous-nonmyeloablative allogeneic transplant
* Chronic lymphocytic leukemia (CLL), non-Hodgkin's lymphoma (NHL) or Hodgkin's Disease (HD) who are ineligible for autologous HSCT or who have resistant/refractory disease and who may benefit from tandem autologous nonmyeloablative allogeneic transplant
* Patients who have received a prior allogeneic HSCT and who have either rejected their grafts or who have become tolerant of their grafts with no active graft-versus-host disease (GvHD) requiring immunosuppressive therapy
* DONOR: Related donors who are identical for one HLA haplotype and mismatched at the HLA-A, -B, -C or DRB1 loci of the unshared haplotype with the exception of single HLA-A, -B or -C allele mismatches

Exclusion Criteria:

* Cross-match positive with donor
* Patients with suitably matched related or unrelated donors
* Patients with conventional transplant options (a conventional transplant should be the priority for eligible patients =< 50 yr of age who have a related donor mismatched for a single HLA-A, -B or DRB1 antigen)
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Presence of active, serious infection (e.g., mucormycosis, uncontrolled aspergillosis, tuberculosis)
* Karnofsky Performance Status < 60 for adult patients
* Lansky-Play Performance Score < 60 for pediatric patients
* Left ventricular ejection fraction < 35%
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 35% and/or receiving supplemental continuous oxygen
* Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL or symptomatic biliary disease
* Human immunodeficiency virus (HIV)-positive patients
* Women of childbearing potential who are pregnant (beta-HCG+) or breast feeding
* Fertile men and women unwilling to use contraceptives during and for 12 months post-transplant
* Life expectancy severely limited by diseases other than malignancy
* DONOR: Donor-recipient pairs in which the HLA-mismatch is only in the HVG direction
* DONOR: Cross-match positive with recipient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Donnell, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data is protected by HIPAA at each participant organization.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nonmyeloablative HSCT): NONMYELOABLATIVE CONDITIONING: Patients receive fludarabine IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 1 hour on days -6 and -5. Patients undergo total body irradiation on day -1.
  TRANSPLANTATION: Patients undergo BMT, from an HLA-haploidentical donor, on day 0.
  POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive cyclophosphamide IV over 1 hour on day 3.
  GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: Patients receive tacrolimus IV over 1-2 hours and then tacrolimus PO, once tolerated, on days 4-180, with taper on day 86 in the absence of graft-versus-host disease. Patients also receive mycophenolate mofetil PO three times daily on days 4-35.
Period: Overall Study
Arm/Group | Treatment (Nonmyeloablative HSCT)
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nonmyeloablative HSCT)
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 40 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 41
  More than one race | 3
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Donor Engraftment (Chimerism)
Description: Defined by the detection of at least 50% donor derived T-cells (CD3+), as a proportion of the total T-cell population
Time Frame: At day +84 after transplantation
Population: Patients receiving haploidentical transplant who had T cell chimerism tested at day +84
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nonmyeloablative HSCT)
Number analyzed (Participants) | 36
Participants | 34

2. Primary Outcome: Incidence of Grades III-IV Acute GVHD
Description: Grade III GVHD represents moderate severity. Grade IV GVHD represents extreme severity
Time Frame: At any time within 200 days after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nonmyeloablative HSCT)
Number analyzed (Participants) | 55
Participants | 4

3. Primary Outcome: Non-relapse-related Mortality
Description: Number of deaths without progression or recurrence of malignant disease
Time Frame: Up to 200 days after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nonmyeloablative HSCT)
Number analyzed (Participants) | 55
Participants | 12

ADVERSE EVENTS:
Arm/Group | Treatment (Nonmyeloablative HSCT)
All-Cause Mortality (participants affected / at risk) | 30/55
Serious Adverse Events (participants affected / at risk) | 11/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nonmyeloablative HSCT) (N=55)
Bacterial infection (Infections and infestations) | 7
Graft-versus-host disease (Immune system disorders) | 2
Secondary myeloid malignancy (Blood and lymphatic system disorders) | 1
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment (Nonmyeloablative HSCT) (N=55)
Invasive Fungal Infection (Infections and infestations) | 6 — Proven or probable invasive fungal infections
CMV reactivation (Infections and infestations) | 27/34
Recurrent or progressive malignancy (Blood and lymphatic system disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes